CLINICAL TRIAL: NCT00780897
Title: Premature Ovarian Failure : Genetic and Physiopathologic Analysis
Brief Title: Premature Ovarian Failure (Genetic and Physiopathologic Analysis)
Acronym: GéNIOP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Myriem Carrier, Department Clinical Research of Developpement
Other Study IDs: P040801
Record Dates: First submitted 2008-10-27; First posted 2008-10-28 (Estimated); Last update posted 2008-10-28 (Estimated); Status verified 2008-10

CONDITIONS: Premature Ovarian Failure
Keywords: PREMATURE OVARIAN FAILURE (POF); GENETIC ANALYSIS; PHYSIOPATHOLOGIC ANALYSIS
MeSH Terms: conditions — Primary Ovarian Insufficiency

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — One ovarian biopsy during the protocol to evaluate ovocytes number and transcriptome analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: POF patients; 18 years <Age> 40 years; Hormonal sampling; FMR1 analysis; FSH Receptor gene analysis; LH Receptor gene analysis; BMP15 gene analysis; GDF9 gene analysis; Connexin 37 analysis; Ovarian biopsy; Bone Mineral Density; Pelvic Ultrasonography;
- 2: Control Group No POF patients; Benign ovarian pathology; 18 years <Age> 40 years; Hormonal sampling; FMR1 analyze; FSH Receptor gene analysis; LH Receptor gene analysis; BMP15 gene analysis; GDF9 gene analysis; Connexin 37 analysis; Ovarian biopsy under specific conditions; Bone Mineral Density; Pelvic Ultrasonography

SUMMARY:
Premature Ovarian Failure (POF), syndrome observed in young woman, present consequences on hormonal and leads at definitive infertility. It's a rare and complex syndrome and for this reason, we propose to initiate a collaborative team network to understand better his genetic and physiopathology.

We are going to realize a global study of this syndrome with clinical and fundamentals approaches. We wish that this project allows us to understand better the physiopathology of this rare disease. Finally, POF responsible genes identification is the base for future development of therapeutics approaches.

DETAILED DESCRIPTION:
Premature ovarian failure (POF) is a rare but not exceptional disease concerning 0.1% of the more-than-thirty-years-old women. On the clinical aspect, patients present a primary or secondary amenorrhea depending on when the disease occurs in their lives. Infertility is most of the time definitive and the yet only available therapy is auto implantation of cryopreserved oocytes. Initiation of a substitutive hormonal treatment is also necessary to prevent the consequences of estrogenic hardship (i.e leading to osteoporosis).

POF has numerous possible origins, and can be linked to auto-immune diseases, metabolic disorders (i.e. galactosemia) or even genetic abnormalities. According to her origin, POF is characterized by (a) a depletion of primary follicles, (b) increased or accelerated follicle atresia (c) an alteration of the recruitment of dominant follicle and (d) stopped follicular maturation.

The purpose of our work is to organize a clinical and fundamental research network focussed on premature ovarian failure (POF). It will aim to collect clinical, biological, radiological and histological information on patients, and according to their phenotypes, to decide for searching possible genetic abnormalities leading to POF. And in the same time, the constitution of a broad tissue collection allows the study of ovarian transcripts, using POF as a pathologic model to describe ovaries and follicle development-involved genes.

ELIGIBILITY:
Inclusion criteria :

Experimental group:

* 18 years <Age> 39 years
* Patient with amenorrhea since at least 3 months
* Patient with at least 1 FSH dosage > 30 mUI/L
* Patients between 40 and 45 years old with hormonal results indicating a POF declared before 39 years old will be included.
* Informed Consent Form Signature

Control group:

* 18 years <Age> 39 years
* Patient having a benign ovarian pathology justifying an ovarian surgery
* Informed Consent Form Signature

Exclusion criteria:

Not applicable

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: POF patients & controls
Sampling Method: Non-Probability Sample
Enrollment: 87 (Estimated)
Dates: Start 2005-03; Primary Completion 2009-03 (Estimated); Study Completion 2009-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Touraine, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Groupe Hopitalier Pitié-Salpêtrière, Paris, France